CLINICAL TRIAL: NCT07163013
Title: Digital Cognitive Behavioral Therapy for Chinese Adolescents With Depressive Symptoms（CADS-D ): A Randomized Clinical Trial
Brief Title: Digital Cognitive Behavioral Therapy for Chinese Adolescents With Depressive Symptoms（CADS-D )
Acronym: CADS-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Zhou, Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1stChongqingMu2
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-09

CONDITIONS: Depressive Symptom
Keywords: Depressive symptoms; Digital cognitive behavioral therapy; Adolescent
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Present study is a single center, two arms, and open-label randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: As the intervention measure set in this study, it is impossible to blind participants or intervention providers. Trained research assistants who are blinded to intervention will conduct the assessment, and data analyst are kept blind to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital cognitive behavioral therapy Group (Experimental): Participants in the intervention group are required to complete two module a week and all modules were be delivered in 6 weeks after the program starts.
  Interventions: Other: Digital cognitive behavioral therapy(DCBT)
- Regular mental health curriculum Group (Other): The participants of control group are allocated to regular mental health curriculum provided by school staff for 6 weeks.
  Interventions: Other: Regular mental health curriculum

INTERVENTIONS:
Other: Digital cognitive behavioral therapy(DCBT) — Moca is a mobile application designed to deliver structural CBT for adolescents with mood problems. Moca provides six-twelve guided sessions with an estimated proceeding duration of 25-45min each, developed to be processed weekly. The content of each session includes the introduction of the core concepts and principles of CBT, psychological counseling dialogue, skill exercises, and homework. Content presentation forms include text, animation, audio, comics, etc. At the end of each module, the participants will be asked to submit homework that will ask them to apply their learned skills to nursing or daily life situations that they personally perceive as stressful. Participants can review the completed sessions and record their mood status during the intervention period.
  Arms: Digital cognitive behavioral therapy Group
Other: Regular mental health curriculum — The content of regular mental health curriculum includes mental health education lecture. Few lectures address the knowledge and skills involved in CBT in such education lecture.
  Arms: Regular mental health curriculum Group

SUMMARY:
CADS-D aimes to evaluate the effectiveness and feasibility of a newly DCBT program for Chinese adolescents with depressive symptoms.

DETAILED DESCRIPTION:
CADS-D is a single-center, two-arm, open-label randomized controlled trial. The trial targeted 12-18 years adolescents with depressive symptoms. Intervention group receives the digital cognitive behavioral therapy (DCBT) program for 6 weeks, while the control group receives the regular mental health curriculum provided by school staff for 6 weeks. Assessments are conducted at three time points: baseline, post-intervention (6 weeks), and at 3 months follow-up (18 weeks). The primary outcome is the effectiveness of DCBT. Secondary outcomes include the feasibility of DCBT, self-reported depressive severity, anxiety severity, psychological resilience, and the quality of life enjoyment and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 to 18 years;
2. Scored 28 or higher on the children's depression rating scale-revised (CDRS-R);
3. Have the ability to read and write in Chinese;
4. Participant and at least one of their guardians provided written consent;
5. Have access to mobile phone and internet.

Exclusion Criteria:

1. The researchers assessed that the adolescent's depressive symptoms were too severe to participate to CADS-D;
2. Scored 5 or higher on item 13 (suicidal ideation) on CDRS-R;
3. Participants who met diagnosis of other mental disorder except depression;
4. Severe physical illnesses or other physical disabilities that prevented the use of DCBT;
5. Within the past three months or currently undergoing any antidepressant treatment, including medication therapy, psychotherapy, and physical therapy;
6. Unavailability to follow up months after intervention.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in CDRS-R (Children's Depression Rating Scale) scores from baseline | Baseline of intervention period, 6 weeks, and 3 months follow-up (18 weeks)
  Children's Depression Rating Scale is a 17 items observer-rated scale developed specifically for children and adolescents. Total scores range from 17-113, with higher scores indicating greater severity of depressive symptoms.

SECONDARY OUTCOMES:
Feasibility of DCBT | 6 weeks
  Feasibility is assessmented by an acceptability and satisfaction questionnaire. The questionnaire constitutes 10 items which designed to examine acceptability and satisfaction with DCBT. In the first 8 questions, participants rated each item on a 5-point Likert scale. In last 2 questions, participants are asked to write the best and worst things about DCBT.
Changes in PHQ (9-item Patient Health Questionnaire) scores from baseline | Baseline of intervention period, 6 weeks, and 3 months follow-up (18 weeks)
  Improvement in self-reported depressive symptoms. Total scores range from 0-27, with higher scores indicating greater severity of self-reported depressive symptoms.
Changes in GAD-7 (Generalized Anxiety Disorder 7-item Scale) scores from baseline | Baseline of intervention period, 6 weeks, and 3 months follow-up (18 weeks)
  Improvement in self-reported anxiety symptom. Total scores range from 0-21, with higher scores indicating greater severity of self-reported anxiety symptoms.
Changes in CD-RISC ( Connor-Davidson Resilience Scale) scores from baseline | Baseline of intervention period, 6 weeks, and 3 months follow-up (18 weeks)
  Improvement in psychological resilience assessed by Connor-Davidson Resilience Scale. Total scores range from 0-100, with higher total scores indicating stronger psychological resilience.
Changes in PQ-LES-Q (The Paediatric Quality of Life Enjoyment and Satisfaction Questionnaire) scores from baseline | Baseline of intervention period, 6 weeks, and 3 months follow-up (18 weeks)
  Improvement of adolescents' quality of life. The total scores range from 14-70，with higher scores indicating greater enjoyment and satisfaction with life.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barker MM, Beresford B, Bland M, Fraser LK. Prevalence and Incidence of Anxiety and Depression Among Children, Adolescents, and Young Adults With Life-Limiting Conditions: A Systematic Review and Meta-analysis. JAMA Pediatr. 2019 Sep 1;173(9):835-844. doi: 10.1001/jamapediatrics.2019.1712. PMID 31282938
- [Background] Janssens KA, Rosmalen JG, Ormel J, van Oort FV, Oldehinkel AJ. Anxiety and depression are risk factors rather than consequences of functional somatic symptoms in a general population of adolescents: the TRAILS study. J Child Psychol Psychiatry. 2010 Mar;51(3):304-12. doi: 10.1111/j.1469-7610.2009.02174.x. Epub 2009 Sep 28. PMID 19788552
- [Background] Pettit JW, Lewinsohn PM, Roberts RE, Seeley JR, Monteith L. The long-term course of depression: development of an empirical index and identification of early adult outcomes. Psychol Med. 2009 Mar;39(3):403-12. doi: 10.1017/S0033291708003851. Epub 2008 Jul 8. PMID 18606049
- [Background] Weissman MM, Wolk S, Goldstein RB, Moreau D, Adams P, Greenwald S, Klier CM, Ryan ND, Dahl RE, Wickramaratne P. Depressed adolescents grown up. JAMA. 1999 May 12;281(18):1707-13. doi: 10.1001/jama.281.18.1707. PMID 10328070
- [Background] O'Keeffe S, Martin P, Goodyer IM, Kelvin R, Dubicka B; IMPACT Consortium; Midgley N. Prognostic Implications for Adolescents With Depression Who Drop Out of Psychological Treatment During a Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2019 Oct;58(10):983-992. doi: 10.1016/j.jaac.2018.11.019. Epub 2019 Apr 1. PMID 30946974
- [Background] Thapar A, Collishaw S, Pine DS, Thapar AK. Depression in adolescence. Lancet. 2012 Mar 17;379(9820):1056-67. doi: 10.1016/S0140-6736(11)60871-4. Epub 2012 Feb 2. PMID 22305766
- [Background] Davey CG, Chanen AM, Hetrick SE, Cotton SM, Ratheesh A, Amminger GP, Koutsogiannis J, Phelan M, Mullen E, Harrison BJ, Rice S, Parker AG, Dean OM, Weller A, Kerr M, Quinn AL, Catania L, Kazantzis N, McGorry PD, Berk M. The addition of fluoxetine to cognitive behavioural therapy for youth depression (YoDA-C): a randomised, double-blind, placebo-controlled, multicentre clinical trial. Lancet Psychiatry. 2019 Sep;6(9):735-744. doi: 10.1016/S2215-0366(19)30215-9. Epub 2019 Jul 29. PMID 31371212
- [Background] Zhou X, Teng T, Zhang Y, Del Giovane C, Furukawa TA, Weisz JR, Li X, Cuijpers P, Coghill D, Xiang Y, Hetrick SE, Leucht S, Qin M, Barth J, Ravindran AV, Yang L, Curry J, Fan L, Silva SG, Cipriani A, Xie P. Comparative efficacy and acceptability of antidepressants, psychotherapies, and their combination for acute treatment of children and adolescents with depressive disorder: a systematic review and network meta-analysis. Lancet Psychiatry. 2020 Jul;7(7):581-601. doi: 10.1016/S2215-0366(20)30137-1. PMID 32563306
- [Background] Fitzpatrick KK, Darcy A, Vierhile M. Delivering Cognitive Behavior Therapy to Young Adults With Symptoms of Depression and Anxiety Using a Fully Automated Conversational Agent (Woebot): A Randomized Controlled Trial. JMIR Ment Health. 2017 Jun 6;4(2):e19. doi: 10.2196/mental.7785. PMID 28588005
- [Background] Rushton J, Bruckman D, Kelleher K. Primary care referral of children with psychosocial problems. Arch Pediatr Adolesc Med. 2002 Jun;156(6):592-8. doi: 10.1001/archpedi.156.6.592. PMID 12038893
- [Background] Ritterband LM, Andersson G, Christensen HM, Carlbring P, Cuijpers P. Directions for the International Society for Research on Internet Interventions (ISRII). J Med Internet Res. 2006 Sep 29;8(3):e23. doi: 10.2196/jmir.8.3.e23. PMID 17032639
- [Background] Imamura K, Kawakami N, Furukawa TA, Matsuyama Y, Shimazu A, Umanodan R, Kawakami S, Kasai K. Does Internet-based cognitive behavioral therapy (iCBT) prevent major depressive episode for workers? A 12-month follow-up of a randomized controlled trial. Psychol Med. 2015 Jul;45(9):1907-17. doi: 10.1017/S0033291714003006. Epub 2015 Jan 7. PMID 25562115
- [Background] Hallgren M, Helgadottir B, Herring MP, Zeebari Z, Lindefors N, Kaldo V, Ojehagen A, Forsell Y. Exercise and internet-based cognitive-behavioural therapy for depression: multicentre randomised controlled trial with 12-month follow-up. Br J Psychiatry. 2016 Nov;209(5):414-420. doi: 10.1192/bjp.bp.115.177576. Epub 2016 Sep 8. PMID 27609813
- [Background] Thase ME, Wright JH, Eells TD, Barrett MS, Wisniewski SR, Balasubramani GK, McCrone P, Brown GK. Improving the Efficiency of Psychotherapy for Depression: Computer-Assisted Versus Standard CBT. Am J Psychiatry. 2018 Mar 1;175(3):242-250. doi: 10.1176/appi.ajp.2017.17010089. Epub 2017 Oct 3. PMID 28969439
- [Background] Kaltenthaler E, Parry G, Beverley C, Ferriter M. Computerised cognitive-behavioural therapy for depression: systematic review. Br J Psychiatry. 2008 Sep;193(3):181-4. doi: 10.1192/bjp.bp.106.025981. PMID 18757972
- [Background] Merry SN, Stasiak K, Shepherd M, Frampton C, Fleming T, Lucassen MF. The effectiveness of SPARX, a computerised self help intervention for adolescents seeking help for depression: randomised controlled non-inferiority trial. BMJ. 2012 Apr 18;344:e2598. doi: 10.1136/bmj.e2598. PMID 22517917
- [Background] Fleming T, Lucassen M, Stasiak K, Sutcliffe K, Merry S. Technology Matters: SPARX - computerised cognitive behavioural therapy for adolescent depression in a game format. Child Adolesc Ment Health. 2021 Feb;26(1):92-94. doi: 10.1111/camh.12444. Epub 2021 Jan 4. PMID 33393723
- [Background] Ivlev I, Beil TL, Haynes JS, Patnode CD. Rapid Evidence Review of Digital Cognitive-Behavioral Therapy for Adolescents With Depression. J Adolesc Health. 2022 Jul;71(1):14-29. doi: 10.1016/j.jadohealth.2022.01.220. Epub 2022 Mar 4. PMID 35256238
- [Background] Yeung A, Wang F, Feng F, Zhang J, Cooper A, Hong L, Wang W, Griffiths K, Bennett K, Bennett A, Alpert J, Fava M. Outcomes of an online computerized cognitive behavioral treatment program for treating chinese patients with depression: A pilot study. Asian J Psychiatr. 2018 Dec;38:102-107. doi: 10.1016/j.ajp.2017.11.007. Epub 2017 Nov 11. PMID 29146042
- [Background] Srivastava P, Mehta M, Sagar R, Ambekar A. Smartteen- a computer assisted cognitive behavior therapy for Indian adolescents with depression- a pilot study. Asian J Psychiatr. 2020 Apr;50:101970. doi: 10.1016/j.ajp.2020.101970. Epub 2020 Feb 19. PMID 32114331